CLINICAL TRIAL: NCT06533904
Title: Percutaneous Cryoablation of Intercostal Nerves for the Treatment of Rib Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 5240003
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Trauma; Rib Fractures; Chest Wall Disorder; Respiratory Insufficiency; Pain, Chest; Rib Trauma; Rib Fracture Multiple; Respiratory Failure; Respiratory Distress Syndrome
Keywords: Trauma; Respiratory Failure; Respiratory Distress; Respiratory Insufficiency; Rib Fractures; Chest Wall Trauma; Percutaneous Cryoablation; Multimodal Pain Therapy; Multimodal Pain Regimen
MeSH Terms: conditions — Wounds and Injuries; Rib Fractures; Respiratory Insufficiency; Chest Pain; Respiratory Distress Syndrome; Dyspnea

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to standard multi-modal pain regimen with percutaneous cryoablation versus standard multi-modal pain regimen alone.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard multi-modal pain regimen alone (Placebo Comparator)
  Interventions: Other: Multi-modal pain regimen
- Standard multi-modal pain regimen with percutaneous cryoablation (Experimental)
  Interventions: Procedure: Percutaneous Cryoablation of Intercostal Nerves; Other: Multi-modal pain regimen

INTERVENTIONS:
Procedure: Percutaneous Cryoablation of Intercostal Nerves — Percutaneous Cryoablation of Intercostal Nerves
  Arms: Standard multi-modal pain regimen with percutaneous cryoablation
Other: Multi-modal pain regimen — Standard rib fracture protocol including cyclooxygenase inhibitors, anti-neuropathic, muscle relaxers, short term anesthesia interventions (percutaneous block, epidural)

SUMMARY:
The goal of this double blinded randomized control trial is to learn if percutaneous cryoablation of traumatic rib fractures improves outcomes. The main questions it aims to answer are:

Does percutaneous cryoablation improve short and long term pain scores? Does percutaneous cryoablation improve short and long term respiratory mechanics? Does percutaneous cryoablation improve long term quality of life? Does percutaneous cryoablation decrease delirium?

Researchers will compare cryoablation to standard multimodal pain therapy to see if this impacts respiratory recovery.

Participants will undergo randomization, percutaneous cryoablative procedure, and participate in tests at pre-determined intervals to evaluate their pulmonary recovery.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* > 2 rib fractures
* Verbal Pain score > 5
* Incentive Spirometry < 60% of predicted

Exclusion Criteria:

* Isolated Fractures of Ribs 1-3 and/or 10-12
* Posterior Rib Fracture < 4 cm from costovertebral joint
* Sternal, Clavicle, Scapula Fracture
* Thoracic Spinal Fracture of any type
* Open Abdominothoracic Surgery
* Unstable Spine
* Extensive Subcutaneous Emphysema
* BMI > 35
* Plan for Rib Plating
* Chronic Opioid Use
* Prior to study enrollment: Intubated, Traumatic Brain Injury, Dementia, Cognitive Impairment, Encephalopathy
* Coagulopathy, Shock at time of ablation
* Inability to participate in activities of daily living prior to injury
* Home O2 use prior to trauma
* Inhalation Injury
* Rib Fractures due to cardiopulmonary resuscitation
* Life Expectancy < 6 months
* > 48 hours from injury
* Pregnant, Incarcerated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Pain Score: Numeric Pain Scale | Through study completion, up to 1 year
  Short and Long Term Pain Scores. Range from 0 to 10 where 0 is no pain and 10 is most severe and worse outcome.
Rate of abnormal respiratory mechanics: Incentive Spirometry | Through study completion, up to 1 year
Rate of abnormal respiratory mechanics: Pulmonary Function Tests | Through study completion, up to 1 year
  Short and Long Term Respiratory Mechanics. Pulmonary Function Tests will specifically measure Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC)
Rate of delirium: Confusion Assessment Method (CAM) Score | Through study completion, up to 1 year
  The score ranges from 0 to 19. Where higher scores indicate more severe delirium and low scores indicate less severe or no delirium
Quality of Life on Survey | Through study completion, up to 1 year
  Long Term Quality of Life

SECONDARY OUTCOMES:
Rate of Pneumonia | Through study completion, up to 1 year
Rate of need for Intubation/Mechanical Ventilation | Through study completion, up to 1 year
Rate of need for tracheostomy | Through study completion, up to 1 year
Number of Ventilatory Days | Through study completion, up to 1 year
ICU Length of Stay | Through study completion, up to 1 year
Hospital Length of Stay | Through study completion, up to 1 year
Acute Respiratory Distress Syndrome | Through study completion, up to 1 year
Rate of Mortality | Through study completion, up to 1 year
Rate of Pleural Space Complications | Through study completion, up to 1 year
  Hemothorax, Delayed hemothorax, Pneumothorax, Empyema, Hydrothorax, Rate of tube thoracostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States